CLINICAL TRIAL: NCT02109653
Title: A Phase II, Single Arm, Open-label, Multicenter, Study of Oral LGX818 in Patients With BRAF V600 Mutant, Advanced Non-small Cell Lung Cancer (NSCLC) That Have Progressed During or After at Least One Prior Chemotherapy
Brief Title: Efficacy and Safety of LGX818 in Patients With Advanced or Metastatic BRAF V600 Mutant NSCLC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never started - transferred to Array.
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLGX818A2202; 2013-005014-34 (EudraCT Number)
Record Dates: First submitted 2014-03-25; First posted 2014-04-10 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC,; Non-Small Cell Lung Cancer,; BRAF V600,; LGX818
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — encorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LGX818 (Experimental): Adult patients, with confirmed diagnosis of BRAF V600E mutant advanced or metastatic NSCLC who have progressed on or after at least one prior systemic anticancer therapy.
  Interventions: Drug: LGX818

INTERVENTIONS:
Drug: LGX818 — Oral LGX818 300mg daily

SUMMARY:
This is an open-label, multi-center, single arm phase II study to evaluate the efficacy and safety of novel BRAF (B-raf murine sarcoma viral oncogene homolog B1) inhibitor encorafenib (LGX818) when used as single agent in patients with advanced or metastatic (stage IIIB or IV) BRAF V600 mutant NSCLC. Patients must have progressed on or after at least one previous systemic, anti-cancer therapy for locally advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Presence of BRAF V600E mutation in tumor tissue
* Histologically or cytologically confirmed diagnosis of Stage IIIB or IV NSCLC
* At least one measurable lesion as defined by RECIST v1.1
* Patients must have progressed during or after at least one previous systemic, anti-cancer treatment for locally advanced or metastatic NSCLC.
* Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance status 0-2

Exclusion Criteria:

* Patients with symptomatic Central Nervous System (CNS) metastases
* History of leptomeningeal metastases
* Prior therapy with a BRAF inhibitor
* Patients taking prohibited medication listed in the protocol
* Presence or history of a malignant disease other than NSCLC that has been diagnosed and/or required therapy within the past 3 years.
* Impaired cardiovascular function or clinically significant cardiovascular diseases
* Pregnant or lactating women or woman of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | up to 24 weeks
  ORR per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 as assessed by investigator

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | baseline, every 6 weeks up to 24 weeks
  ORR per RECIST 1.1 as assessed by by Blinded independent review committee (BIRC)
Progression-Free Survival (PFS) | baseline, every 6 weeks up to 24 weeks
  PFS determined by investigator and BIRC.
Duration of Response (DOR) | baseline, every 6 weeks up to 24 weeks
  DOR by investigator and BIRC assessments.
Overall survival (OS) | baseline, every 6 weeks up to 24 weeks
  Overall survival (OS)
Safety Profile | baseline, every 3 weeks up to 24 weeks
  Adverse events and laboratory abnormalities
Disease Control Rate (DCR) | baseline, every 6 weeks up to 24 weeks
  DCR by investigator and BIRC assessments.
Pharmacokinetics profile | baseline, every 3 weeks up to 18 weeks
  Plasma concentration-time profiles of encorafenib (LGX818).
Concordance between the BRAF mutation status from investigational diagnostic test and the companion diagnostic assay | screening, up to 24 weeks
  Concordance rate between BRAF mutation status obtained using the investigational diagnostic test and the companion diagnostic assay which will be submitted for Pre-market approval (PMA)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — 1-800-718-1021
Locations (1):
- University of Chicago Medical Center SC-2, Chicago, Illinois, United States